CLINICAL TRIAL: NCT00093210
Title: A Double-Blind, Randomized, Crossover Evaluation of the Pharmacokinetics of Recombinant Human Factor IX (BeneFIX) and a New Formulation of BeneFIX (rFIX-R); and an Open-Label Safety and Efficacy Evaluation of rFIX-R in Previously Treated Patients With Moderate to Severe (FIX:C≤2%) Hemophilia B
Brief Title: Study Evaluating of Recombinant Human Factor IX (BeneFIX) and a New Formulation of BeneFIX (rFIX-R) in Moderate to Severe Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 3090A1-304
Record Dates: First submitted 2004-10-04; First posted 2004-10-07 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

INTERVENTIONS:
Drug: rFIX
Drug: rFIX-R

SUMMARY:
The primary objective of this clinical research study is to establish the bioequivalence of 2 treatments, rFIX and rFIX-R, when given as a 10-minute intravenous bolus infusion.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe hemophilia B (FIX: C ≤2%)
* Previously treated patients (PTPs) with ≥150 documented exposure days
* Age ≥ 12 years (US sites only)

Exclusion Criteria:

* Detectable factor IX inhibitor defined as ≥0.6 Bethesda Units for pooled plasma reported by the local laboratory (family history of inhibitors will not exclude the patient)
* Patient history of factor IX inhibitor replacement therapy
* Patient unable to be off factor IX replacement therapy for at least 5 days without bleeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Rendo P, Smith L, Lee HY, Shafer F. Nonacog alfa: an analysis of safety data from six prospective clinical studies in different patient populations with haemophilia B treated with different therapeutic modalities. Blood Coagul Fibrinolysis. 2015 Dec;26(8):912-8. doi: 10.1097/MBC.0000000000000359. PMID 26196195